CLINICAL TRIAL: NCT01475838
Title: A Phase 3b Randomized, Open-Label Study to Evaluate Switching From Regimens Consisting of a Ritonavir-boosted Protease Inhibitor (PI + RTV) Plus Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) to the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate Single-Tablet Regimen (EVG/COBI/FTC/TDF) in Virologically-Suppressed, HIV-1 Infected Patients
Brief Title: Study to Evaluate Switching From Regimens Consisting of a Ritonavir-boosted Protease Inhibitor Plus Emtricitabine/Tenofovir Fixed-Dose Combination to the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir DF Single-Tablet Regimen in Virologically Suppressed, HIV-1 Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-236-0115; 2011-004483-30 (EudraCT Number)
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; HIV; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stribild (Experimental): Participants will switch from their baseline treatment regimen to Stribild for up to 96 weeks, and may continue to receive Stribild in the extension phase.
  Interventions: Drug: Stribild
- PI+RTV+FTC/TDF (Active Comparator): Participants will stay on their baseline treatment regimen antiretroviral regimen consisting of a PI boosted with RTV plus FTC/TDF for up to 96 weeks, and may switch to Stribild in the extension phase.
  Interventions: Drug: PI; Drug: RTV; Drug: FTC/TDF; Drug: Stribild

INTERVENTIONS:
Drug: PI — PI administered according to prescribing information; allowed PIs include atazanavir (ATV), darunavir (DRV), fosamprenavir (FPV), lopinavir (LPV), or saquinavir (SQV)
  Arms: PI+RTV+FTC/TDF
Drug: RTV — RTV administered according to prescribing information FTC/TDF administered according to prescribing information
  Arms: PI+RTV+FTC/TDF
Drug: FTC/TDF — FTC/TDF (200/300 mg) administered according to prescribing information
  Other Names: Truvada
  Arms: PI+RTV+FTC/TDF
Drug: Stribild — Stribild (E/C/F/TDF) (150/150/200/300 mg) STR administered orally once daily with food

SUMMARY:
This study will evaluate the non-inferiority of Stribild® (elvitegravir/cobicistat/ emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF)) single-tablet regimen (STR) relative to regimens consisting of a protease inhibitor (PI) boosted with ritonavir (RTV) plus Truvada® (FTC/TDF) fixed-dose combination in maintaining HIV-1 RNA < 50 copies/mL at Week 48 in virologically suppressed, HIV-1 infected adults. This study will also evaluate the safety, tolerability, and efficacy of the two regimens through 96 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Be on a stable antiretroviral regimen consisting of a ritonavir boosted PI plus FTC/TDF continuously for ≥ 6 consecutive months preceding the screening visit
* Be on the first or second antiretroviral drug regimen documented undetectable plasma HIV 1 RNA levels for ≥ 6 months preceding the screening visit
* No previous use of any approved or experimental integrase strand transfer inhibitor (INSTI) for any length of time
* Documented historical genotype prior to starting initial antiretroviral therapy showing no known resistance to TDF or FTC
* HIV RNA < 50 copies/mL at screening
* Normal ECG
* Hepatic transaminases ≤ 5 × the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Estimated glomerular filtration rate ≥ 70 mL/min
* Females of childbearing potential must agree to utilize highly effective contraception methods, or be nonheterosexually active, practice sexual abstinence from screening throughout the duration of the study period and for 30 days following the last dose of study drug
* Female participants who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Male participants must agree to utilize a highly effective method of contraception during heterosexual intercourse from the screening visit, throughout the duration of the study and for 30 days following discontinuation of investigational medicinal product, or must be nonheterosexually active, or practice sexual abstinence
* Age ≥ 18 years

Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Receiving drug treatment for hepatitis C, or participants who are anticipated to receive treatment for hepatitis C during the course of the study
* Experiencing decompensated cirrhosis
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance abuse that would interfere with compliance
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 30 days prior to Baseline, except for intramuscular penicillin for the treatment of syphilis
* Have been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study
* Receiving ongoing therapy with any of the medications, including drugs not to be used with elvitegravir, cobicistat, FTC, or TDF; or those with any known allergies to the excipients of E/C/F/TDF tablets, or FTC/TDF tablets
* No anticipated need to initiate drugs during the study that are contraindicated
* Receiving other investigational drugs
* Participation in any other clinical trial
* Any other clinical condition or prior therapy that would make the participant unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thai Nguyen-Cleary, Study Director — Gilead Sciences
Locations (99):
- United States (45):
  - Spectrum Medical Group, Phoenix, Arizona
  - Pueblo Family Physicians, Phoenix, Arizona
  - AIDS Healthcare Foundation, Beverly Hills, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Kaiser Permanente, Hayward, California
  - Kaiser Permanente, Los Angeles, California
  - Peter J. Ruane, M.D., Inc., Los Angeles, California
  - OASIS Clinic, Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Kaiser Permanente, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Dupont Circle Physicians Group, P.C, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Gary Richmond, MD, Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Idocf/Valuhealthmd, Llc, Orlando, Florida
  - Infectious Diseases Associates of NW FL, P.A., Pensacola, Florida
  - AHF Health Positive Tampa Bay, Safety Harbor, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - Northwestern University Division of Infectious Diseases, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County/Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Be Well Medical Center, Berkley, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - The Kansas City Free Health Clinic, Kansas City, Missouri
  - I.D. Care Associates PA, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Greiger Clinic, Mount Vernon, New York
  - ID Consultants, P.A., Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Uptown Physicians Group, Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon Crofoot Md, Pa, Houston, Texas
  - St. Hope Foundation Inc, Houston, Texas
- Austria (4):
  - Innsbruck Medical University, Innsbruck
  - Univ.-Kklinik fuer Innere Medizin III, Salzburg
  - Medical University of Vienna, Vienna
  - Otto-Wagner-Spital, Vienna
- Belgium (3):
  - UCL Saint Luc, Brussels
  - University Hospital Ghent, Ghent
  - CHU Sart Tilman, Liège
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique Medicale Du Quartier Latin, Montreal, Quebec
- France (10):
  - CHU de Besancon, Hopital Saint-Jacques, Besançon
  - Hôpital de la Croix-Rousse, Lyon
  - CHU Hôpital Gui de Chauliac, Montpellier
  - Archet 1 Chu Nice Department of Infectology, Nice
  - Saint-Louis Hospital, Paris
  - Hopital Saint Antoine, Paris
  - Hôpital Bichat-Claude Bernard, Paris
  - hôpital Tenon, Paris
  - Maladies Infectieuses Dpt, Paris
  - Hôpital Haut Lévêque, Pessac
- Germany (9):
  - Epimed GmbH, Berlin
  - University of Bonn, Bonn
  - Infektlonsambulanz Unlkllnik Koln, Cologne
  - Universitätsklinikum Essen, Dermatologie, HIV Ambulanz, Essen
  - Johann Wolfgang Goethe-University Hospital / Infectious Diseases Hs 68, Frankfurt
  - ICH Study Center, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Ambulanzzentrum des UKE GmbH, Bereich Infektiologie, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Infektionsambulanz, Med Poliklink, Klinikum der Universitat Munchnen, Munich
- Italy (6):
  - Ospedali Riuniti, Bergamo
  - Fondazione Centro San Raffaele, Milan
  - Clinic of Infectious Diseases, University of Milan-San Paolo Hospital, Milan
  - Ospedale Luigi Sacco, Milan
  - National Institute for Infectious Diseases "L. Spallanzani", Rome
  - University of Torino, Dept of Infectious Disease, Torino
- Portugal (3):
  - HHP Hospital de Cascais, Alcabideche
  - Hospital de Santa Maria-CHLN, EPE, Lisbon
  - Hospital Santo Antonio Dos Capuchos, Centro Hospitalar de Lisboa, Lisbon
- Puerto Rico (2):
  - Clinical Research Puert Rico, San Juan
  - University of Puerto Rico School of Medicine, San Juan
- Spain (9):
  - Hospital General Universitario Alicante, Alicante
  - Hospital clinic, Barcelona
  - Hospital Universitari Bellvitge HIV Unit. Infectious Disease Service., Barcelona
  - Hospital Germans Trias I Pujol, Barcelona
  - Hospital General Universitario de Elche, Elche, Alicante
  - Infectious Diseases Department, Hospital Carlos III, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Hospital Virgen del Rocio, Seville
- Switzerland (3):
  - Geneva University Hospital, Geneva
  - University Hospital of Zurich; Division of Infectious Diseases and Hospital Epidemiology, Zurich
  - Zentrum fur Infektionskrankheiten, Zurich
- United Kingdom (3):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Royal Free Hampstead NHS Trust, London
  - Chelsea and Westminster, London

REFERENCES:
- [Result] Arribas JR, Pialoux G, Gathe J, Di Perri G, Reynes J, Tebas P, Nguyen T, Ebrahimi R, White K, Piontkowsky D. Simplification to coformulated elvitegravir, cobicistat, emtricitabine, and tenofovir versus continuation of ritonavir-boosted protease inhibitor with emtricitabine and tenofovir in adults with virologically suppressed HIV (STRATEGY-PI): 48 week results of a randomised, open-label, phase 3b, non-inferiority trial. Lancet Infect Dis. 2014 Jul;14(7):581-9. doi: 10.1016/S1473-3099(14)70782-0. Epub 2014 Jun 5. PMID 24908551
- [Result] Pozniak A, Markowitz M, Mills A, Stellbrink HJ, Antela A, Domingo P, Girard PM, Henry K, Nguyen T, Piontkowsky D, Garner W, White K, Guyer B. Switching to coformulated elvitegravir, cobicistat, emtricitabine, and tenofovir versus continuation of non-nucleoside reverse transcriptase inhibitor with emtricitabine and tenofovir in virologically suppressed adults with HIV (STRATEGY-NNRTI): 48 week results of a randomised, open-label, phase 3b non-inferiority trial. Lancet Infect Dis. 2014 Jul;14(7):590-9. doi: 10.1016/S1473-3099(14)70796-0. Epub 2014 Jun 5. PMID 24908550
- [Derived] Arribas JR, DeJesus E, van Lunzen J, Zurawski C, Doroana M, Towner W, Lazzarin A, Nelson M, McColl D, Andreatta K, Swamy R, Szwarcberg J, Nguyen T. Simplification to single-tablet regimen of elvitegravir, cobicistat, emtricitabine, tenofovir DF from multi-tablet ritonavir-boosted protease inhibitor plus coformulated emtricitabine and tenofovir DF regimens: week 96 results of STRATEGY-PI. HIV Clin Trials. 2017 May;18(3):118-125. doi: 10.1080/15284336.2017.1330440. Epub 2017 May 30. PMID 28555519
- [Derived] Gathe J, Arribas JR, Van Lunzen J, Garner W, Speck RM, Bender R, Shreay S, Nguyen T. Patient-Reported Symptoms over 48 Weeks in a Randomized, Open-Label, Phase 3b Non-inferiority Trial of Adults with HIV Switching to Coformulated Elvitegravir, Cobicistat, Emtricitabine, and Tenofovir DF Versus Continuation of Ritonavir-Boosted Protease Inhibitor with Emtricitabine and Tenofovir DF. Patient. 2015 Oct;8(5):445-54. doi: 10.1007/s40271-015-0137-9. PMID 26286337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 18 November 2011. The last study visit occurred on 09 December 2014
Pre-assignment Details: 632 participants were screened.
Groups:
- Stribild: Participants switched from their baseline treatment regimen to Stribild® (elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate; E/C/F/TDF) (150/150/200/300 mg) single-tablet regimen (STR) once daily for up to 96 weeks in the randomized phase, and may have continued to receive Stribild in the extension phase.
- PI+RTV+FTC/TDF: Participants stayed on their baseline treatment regimen consisting of a protease inhibitor (PI) (atazanavir (ATV), darunavir (DRV), fosamprenavir (FPV), lopinavir (LPV), or saquinavir (SQV)) boosted with ritonavir (RTV) plus emtricitabine (FTC)/TDF (200/300 mg) (administered according to prescribing information) for up to 96 weeks in the randomized phase, and may have switched to Stribild in the extension phase.
Period: Randomized Phase
Arm/Group | Stribild | PI+RTV+FTC/TDF
Started | 293 | 145
Completed | 263 | 109
Not Completed | 30 | 36
Not completed — Randomized but Not Treated | 0 | 5
Not completed — Adverse Event | 6 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Investigators Discretion | 1 | 2
Not completed — Withdrew Consent | 10 | 14
Not completed — Lost to Follow-up | 3 | 4
Not completed — Participant Noncompliance | 1 | 5
Not completed — Protocol Violation | 9 | 4
Period: Extension Phase
Arm/Group | Stribild | PI+RTV+FTC/TDF
Started | 42 | 20
Completed | 41 | 20
Not Completed | 1 | 0
Not completed — Participant Noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study medication.
Groups:
- Stribild: Participants switched from their baseline treatment regimen to Stribild (E/C/F/TDF) (150/150/200/300 mg) STR once daily for up to 96 weeks in the randomized phase, and may have continued to receive Stribild in the extension phase.
- PI+RTV+FTC/TDF: Participants stayed on their baseline treatment regimen consisting of a PI (ATV, DRV, FPV, LPV, or SQV) boosted with RTV plus FTC/TDF (200/300 mg) (administered according to prescribing information) for up to 96 weeks in the randomized phase, and may have switched to Stribild in the extension phase.
- Total: Total of all reporting groups
Arm/Group | Stribild | PI+RTV+FTC/TDF | Total
Number analyzed (Participants) | 293 | 140 | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9.7) | 41 (8.9) | 41 (9.4)
Age, Customized [Number; unit: participants]
  < 40 years | 130 | 68 | 198
  ≥ 40 to < 50 years | 109 | 49 | 158
  ≥ 50 years | 54 | 23 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 19 | 62
  Male | 250 | 121 | 371
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 7 | 2 | 9
  Black or African Heritage | 43 | 20 | 63
  White | 234 | 113 | 347
  Other | 5 | 2 | 7
  Not Permitted | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 42 | 17 | 59
  Non-Hispanic/Latino | 249 | 123 | 372
  Not Permitted | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Portugal | 12 | 7 | 19
  France | 39 | 15 | 54
  United States | 84 | 40 | 124
  Puerto Rico | 3 | 2 | 5
  Canada | 5 | 3 | 8
  Spain | 28 | 21 | 49
  Belgium | 6 | 2 | 8
  Austria | 11 | 4 | 15
  Germany | 36 | 21 | 57
  United Kingdom | 13 | 1 | 14
  Switzerland | 12 | 8 | 20
  Italy | 44 | 16 | 60
HIV-1 RNA Category [Number; unit: participants]
  < 50 copies/mL | 291 | 137 | 428
  50 to < 200 copies/mL | 2 | 2 | 4
  200 to < 400 copies/mL | 0 | 0 | 0
  ≥ 400 copies/mL | 0 | 1 | 1
CD4+ Cell Count [Mean (Standard Deviation); unit: cells/µL] | 604 (274.6) | 624 (269.9) | 610 (272.9)
CD4+ Cell Count Category [Number; unit: participants]
  ≤ 50 cells/µL | 0 | 0 | 0
  51 to ≤ 200 cells/µL | 9 | 6 | 15
  201 to ≤ 350 cells/µL | 37 | 14 | 51
  351 to ≤ 500 cells/µL | 69 | 26 | 95
  > 500 cells/µL | 178 | 94 | 272
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 214 | 105 | 319
  Symptomatic HIV Infections | 38 | 17 | 55
  AIDS | 41 | 18 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The FDA-defined Snapshot algorithm was used, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time.
Time Frame: Week 48
Population: Full Analysis Set: Participants who were randomized and treated, and had no major eligibility criteria violations
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | PI+RTV+FTC/TDF
Number analyzed (Participants) | 290 | 139
percentage of participants | 93.8 | 87.1
Statistical Analysis 1: Comparison: Stribild vs PI+RTV+FTC/TDF; Test type: Non-Inferiority or Equivalence — The null hypothesis was that the Stribild group was at least 12% worse than the PI+RTV+FTC/TDF group with respect to the percentage of participants maintaining HIV-1 RNA < 50 copies/mL at Week 48. The alternative hypothesis was that the Stribild group was less than 12% worse than the PI+RTV+FTC/TDF group; p = 0.025, Fisher Exact; Difference in proportions = 6.7, 95% CI 2-sided [0.4 to 13.7] — The 95% confidence interval (CI) for the difference was from unconditional exact method using 2 inverted 1-sided tests with the standardized statistic using StatXact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Description: as for outcome 1
Time Frame: Week 96
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | PI+RTV+FTC/TDF
Number analyzed (Participants) | 290 | 139
percentage of participants | 86.9 | 69.8

3. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed; the missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | PI+RTV+FTC/TDF
Number analyzed (Participants) | 270 | 120
cells/µL | 40 (169.5) | 32 (166.1)

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with available data while on study drug were analyzed; the missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | PI+RTV+FTC/TDF
Number analyzed (Participants) | 255 | 104
cells/µL | 61 (196.5) | 71 (173.4)

ADVERSE EVENTS:
Time Frame: Baseline through end of study (average 88 weeks)
Description: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug
Groups:
- Stribild: Adverse events for this reporting group include those occurring in participants receiving Stribild in the randomized phase.
  Participants switched from their baseline treatment regimen to Stribild (E/C/F/TDF) (150/150/200/300 mg) STR once daily for up to 96 weeks in the randomized phase, and may have continued to receive Stribild in the extension phase.
- PI+RTV+FTC/TDF: Adverse events for this reporting group include those occurring in participants receiving PI+RTV+FTC/TDF in the randomized phase.
  Participants stayed on their baseline treatment regimen consisting of a PI (ATV, DRV, FPV, LPV, or SQV) boosted with RTV plus FTC/TDF (200/300 mg) (administered according to prescribing information) for up to 96 weeks in the randomized phase, and may have switched to Stribild in the extension phase.
- All Stribild: Adverse events for this reporting group include those occurring in participants while receiving Stribild in the randomized and extension phases.
Arm/Group | Stribild | PI+RTV+FTC/TDF | All Stribild
Serious Adverse Events (participants affected / at risk) | 24/293 | 11/140 | 24/313
Other Adverse Events (participants affected / at risk) | 169/293 | 67/140 | 169/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=293) | PI+RTV+FTC/TDF (N=140) | All Stribild (N=313)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 1
Penile abscess (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 2
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=293) | PI+RTV+FTC/TDF (N=140) | All Stribild (N=313)
Diarrhoea (Gastrointestinal disorders) | 27 | 11 | 27
Nausea (Gastrointestinal disorders) | 22 | 5 | 22
Gastroenteritis (Infections and infestations) | 11 | 7 | 11
Nasopharyngitis (Infections and infestations) | 39 | 20 | 39
Pharyngitis (Infections and infestations) | 16 | 7 | 16
Sinusitis (Infections and infestations) | 15 | 6 | 16
Syphilis (Infections and infestations) | 20 | 6 | 20
Upper respiratory tract infection (Infections and infestations) | 29 | 8 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 4 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 4 | 24
Headache (Nervous system disorders) | 24 | 10 | 24
Anxiety (Psychiatric disorders) | 19 | 5 | 20
Depression (Psychiatric disorders) | 18 | 9 | 18
Insomnia (Psychiatric disorders) | 13 | 8 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 6 | 20

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years